CLINICAL TRIAL: NCT04461873
Title: The Effect of Reiki on the Stress Level of Caregivers of Cancer Patients: Qualitative and Single-blind Randomized Controlled Trial
Brief Title: The Effect of Reiki on the Stress Level of Caregivers of Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ulviye ÖZCAN YÜCE, Lecturer doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TDK-2018-8030
Record Dates: First submitted 2020-06-28; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Caregiver Stress Syndrome; Reiki; Caregiver Burnout
Keywords: Care; Stress; Reiki; Nursing
MeSH Terms: conditions — Caregiver Burden | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: The study was conducted using a pre-test and post-test, single-blind randomized controlled trial pattern and semi-structured in-depth interview method of qualitative research.
Who Masked: Participant
Masking Description: The patients of the caregivers who met the study criteria were listed according to the protocol numbers and the participants were assigned to the reiki and sham reiki groups using simple random sampling method by the charge nurse of the chemotherapy unit. Thus, the participants were blinded to the intervention and placebo groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki (Experimental): Reiki was applied to this arm by the researcher who completed her second level education according to the Usui method, for 45 minutes once a week for 6 weeks and by touching the 9 main points in line. A saliva sample was taken from the participants in order to determine the stress level through cortisol and Caregiver Stress Scale (CSS) was applied in the first week of Reiki application. Systolic and diastolic blood pressures and pulse rates were measured for six weeks before and after each application. At the end of six weeks, saliva samples were collected and CSS was applied again. After the 6-week Reiki application, all the caregivers of the intervention group were asked about their experience and opinions regarding the application by the individual in-depth interview method during the home visit.
  Interventions: Other: Reiki
- Sham Reiki (Placebo Comparator): Four student nurses who did not receive Reiki training and were trained about application by the investigator applied sham by gesturing and mimic imitation through touching 9 points for 45 minutes/week for 6 weeks in line. A saliva sample was taken from the participants in order to determine the stress level through cortisol and Caregiver Stress Scale (CSS) was applied in the first week of Reiki application. Systolic and diastolic blood pressures and pulse rates were measured for six weeks before and after each application. At the end of six weeks, saliva samples were collected and CSS was applied again.
  Interventions: Other: Sham Reiki

INTERVENTIONS:
Other: Reiki — Reiki by touching
  Arms: Reiki
Other: Sham Reiki — Sham reiki by gesturing and mimic imitation through touching
  Arms: Sham Reiki

SUMMARY:
Stress caused by late-identified and unmet needs of caregivers negatively affect the physical and emotional health of patients and caregivers as well as their compliance with the treatment. Therefore, it is necessary to evaluate the problems experienced by caregivers and to plan a number of attempts to reduce stress levels. Complementary and integrated practices for caregivers to manage their stresses are increasingly preferred approaches in recent years for many different reasons. One of these integrative practices, Reiki, is an energy therapy involving the use of energy that flows naturally from the hands of the practitioner to strengthen the body's ability to heal itself in order to increase well-being. This study was conducted using a pre-test and post-test, single-blind randomized controlled trial pattern and semi-structured in-depth interview method of qualitative research in order to evaluate the effect of Reiki on stress levels applied to individuals caring for cancer patients. The study comprised 42 women who were primary caregivers of cancer patients in total, as 21 women in Reiki group and 21 women in sham Reiki group. The approval of ethics committee, permissions from the institutions, and informed voluntary approval of the individuals were obtained to conduct the research. The data of the research were collected through the application of Caregiver Stress Scale (CSS), form for care giver's opinions on Reiki experience and application monitoring form including cortisol levels analyzed from saliva samples collected before and after application and measurements of pulse rate and blood pressure values. While Reiki group received reiki to 9 main points for 45 minutes per day for 6 weeks, in the sham Reiki group the same points were touched during the same period without starting energy flow. Caregiver Stress Scale (CSS) and salivary cortisol level were evaluated at the baseline and end of the study, whereas systolic and diastolic blood pressure and pulse rate were evaluated before and after application every week. At the end of the study, the opinions of the Reiki group on Reiki experience were collected by using a form consisting of semi-structured questions. The value of p<0.05 was accepted statistically significant in the data analyses. Descriptive and content analysis methods were used to evaluate the qualitative data.

DETAILED DESCRIPTION:
In this study, women who care for cancer patients received reiki to 9 main points including 7 chakra as well as ankle and feet for 45 minutes once a week for 6 weeks to determine its effect on stress level using a pretest-posttest randomized controlled single-blind study design of quantitative trial and semi-structured in-depth interview method of qualitative trial.The study was conducted in the medical oncology unit of a university hospital in Turkey. The data collection process continued from August 2018 to April 2019 and was reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. To be included in the study, a total of 86 caregivers were directed to the investigator by the charge nurse of the chemotherapy unit. The investigator evaluated the criteria for inclusion into study by conducting a preliminary interview with the directed caregivers. A total of 86 caregivers were evaluated; 61 were found eligible for the study and 51 caregivers agreed to participate into the study. Caregivers were assigned to reiki and sham reiki groups. One caregiver in the Reiki group was excluded from the study on the first application day because he/she could not provide a saliva sample. 4 of the caregivers in the sham reiki group did not continue their application appointments after the first week, and 4 of the caregivers in the sham reiki group left the study stating that they did not want to continue due to the deterioration in prognosis of the caretakers. The study was completed with a total of 42 caregivers

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old and female
* Can communicate
* Being a primary caregiver family member of cancer patients receiving treatment,
* Providing care to the patient for 8 hours / day for at least 6 months, and Caregiver Stress Scale (CSS) score of 7 and above

Exclusion Criteria:

* To provide maintenance service for a fee,
* Having another medical problem that will prevent pulse rate and blood pressure measurement,
* Pulse rate to be variable,
* Being unable to give a saliva secretion due to other medical problems,
* Using cortisol and its derivative drugs,
* Having a history of psychiatric disorders,
* Being a Reiki practitioner or trainer,
* To have received energy therapies such as Reiki / Therapeutic touch / Healing touch,
* To use other complementary and integrated medicine applications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Considering the privacy concerns that the reiki, which is applied by touch, can cause the participants, it is preferred that the participants are women like the practitioners.
Enrollment: 42 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-04-06 (Actual)

PRIMARY OUTCOMES:
Caregiver Stress Scale (CSS) | Change from baseline score at the end of the sixth week
  The Caregiver Stress Scale (CSS) was developed by Robinson (1983) and is a tool that can be used to quickly identify families with potential care concerns. The scale consists of 13 items, which are answered "yes", "no". The main issues are job status, financial situation, physical condition, social status and time. The lowest score that can be obtained from the scale is "0" and the highest score is "13". The positive response to 7 or more items on the scale (7 points and above) indicates that stress is perceived high by the caregiver. In his study, Robinson has obtained a cronbach alpha value of 0.86. Validity and reliability of the Turkish version of the scale was performed by Uğur (2006) and the cronbach alpha value of the scale was calculated as 0.75.
Evaluation of Saliva Cortisol | Change from baseline score at the end of the sixth week
  Saliva samples were collected by a saliva cortisol tube, the amount of cortisol in saliva was measured by electrochemiluminescence immunological test (ECLIA) method using a specific device in the external laboratory. Taking into account that the production of peak cortisol is early in the morning, the samples were collected between 06:00 and 10:00, the reference value for this time interval is <0.874 ug/dL
Application Monitoring Form for Blood Pressure | Change from before and after each application and from the first week to the sixth week
  It includes stimuli of the sympathetic nervous system, such as physiological stress response to emotional stress, high blood pressure and increased pulse rate. Studies show that reiki stimulates parasympathetic activity and balances systolic and diastolic blood pressure and pulse rate. In the light of this information in this study blood pressure (systolic and diastolic blood pressure in mmHg) measurements performed before and after each application were measured three times at five-minute intervals and the mean value of three measurements recorded to minimize variations between measurements.
Application Monitoring Form for Pulse Rate | Change from before and after each application and from the first week to the sixth week
  In order to reveal the retarding effects of Reiki on the pulse rate, similar to its effects on blood pressure, the pulse rate (beats per min) of individuals was measured three times at five-minute intervals and the average value of three measurements was recorded to minimize differences between measurements.
Form for Care Giver's Opinions on Reiki Experience | At the end of the sixth week of Reiki intervation
  It was created in line with the literature in order to get the experience and opinions of the individuals after Reiki application in the reiki group by the individual in-depth interview method. In this form, there are semi-structured questions under the titles of caregivers' "thoughts on the reiki application", "thoughts on the application of reiki to patients they care for in order to reduce the stress level", "thoughts on the application of reiki by the nurses to patients they care for during their hospitalization". While the questions in the form were being structured, the investigator consulted an expert on sociology regarding the themes created from the given answers and the integrity of the expression.

CONTACTS AND LOCATIONS:
Overall Officials: Ulviye Özcan Yüce, Principal Investigator — Osmaniye Korkut Ata Üniversitesi
Locations (1):
- Osmaniye Korkut Ata University, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akmansu M. Integrative oncology. Turk J Oncology. 2019;34(1):56-58.
- [Background] Buckley TM, Schatzberg AF. On the interactions of the hypothalamic-pituitary-adrenal (HPA) axis and sleep: normal HPA axis activity and circadian rhythm, exemplary sleep disorders. J Clin Endocrinol Metab. 2005 May;90(5):3106-14. doi: 10.1210/jc.2004-1056. Epub 2005 Feb 22. PMID 15728214
- [Background] Cassidy N, Collins K, Cyr D, Magni K. The effect of Reiki on women's preoperative anxiety in an ambulatory surgery center. Journal of PeriAnesthesia Nursing, 2010; 25 (3): 196-198.
- [Background] Chang HY, Chiou CJ, Chen NS. Impact of mental health and caregiver burden on family caregivers' physical health. Arch Gerontol Geriatr. 2010 May-Jun;50(3):267-71. doi: 10.1016/j.archger.2009.04.006. Epub 2009 May 13. PMID 19443058
- [Background] Dissiz G, Yilmaz M. Complementary and alternative therapies and health literacy in cancer patients. Complement Ther Clin Pract. 2016 May;23:34-9. doi: 10.1016/j.ctcp.2016.02.004. Epub 2016 Mar 2. PMID 27157956
- [Background] Friedman RS, Burg MM, Miles P, Lee F, Lampert R. Effects of Reiki on autonomic activity early after acute coronary syndrome. J Am Coll Cardiol. 2010 Sep 14;56(12):995-6. doi: 10.1016/j.jacc.2010.03.082. No abstract available. PMID 20828654
- [Background] Lopez G, Mao JJ, Cohen L. Integrative Oncology. Med Clin North Am. 2017 Sep;101(5):977-985. doi: 10.1016/j.mcna.2017.04.011. Epub 2017 Jun 23. PMID 28802474
- [Background] Mackay N, Hansen S, McFarlane O. Autonomic nervous system changes during Reiki treatment: a preliminary study. J Altern Complement Med. 2004 Dec;10(6):1077-81. doi: 10.1089/acm.2004.10.1077. PMID 15674004
- [Background] Musal N. Applied reiki handbook for first degree. İstanbul:Akis Yayıncılık; 2008.
- [Background] Olson K, Hanson J, Michaud M. A phase II trial of Reiki for the management of pain in advanced cancer patients. J Pain Symptom Manage. 2003 Nov;26(5):990-7. doi: 10.1016/s0885-3924(03)00334-8. PMID 14585550
- [Background] Salles LF, Vannucci L, Salles A, Silva MJP. The effect of Reiki on blood hypertension. Acta Paul Enferm. 2014; 27(5):479-84.
- [Background] Tekin HH. In-depth interview of qualitative research method as a data collection technique. İstanbul Üniversitesi Sosyoloji Dergisi 2006;3(13): 101 - 116.
- [Background] Tsigos C, Chrousos GP. Hypothalamic-pituitary-adrenal axis, neuroendocrine factors and stress. J Psychosom Res. 2002 Oct;53(4):865-71. doi: 10.1016/s0022-3999(02)00429-4. PMID 12377295
- [Background] Uğur Ö. Examination of care burden of caregivers of oncology patients. Ege University: Health Sciences Institute, Ph.D. Thesis, İzmir: 2006
- [Background] Vogeser M, Kratzsch J, Ju Bae Y, Bruegel M, Ceglarek U, Fiers T, Gaudl A, Kurka H, Milczynski C, Prat Knoll C, Suhr AC, Teupser D, Zahn I, Ostlund RE. Multicenter performance evaluation of a second generation cortisol assay. Clin Chem Lab Med. 2017 May 1;55(6):826-835. doi: 10.1515/cclm-2016-0400. PMID 27898397
- [Background] Witt CM, Balneaves LG, Cardoso MJ, Cohen L, Greenlee H, Johnstone P, Kucuk O, Mailman J, Mao JJ. A Comprehensive Definition for Integrative Oncology. J Natl Cancer Inst Monogr. 2017 Nov 1;2017(52). doi: 10.1093/jncimonographs/lgx012. PMID 29140493
- [Background] Yıldız E, Dedeli Ö, Pakyüz SÇ. Evaluation of Care Burden and Quality of Life among Family Caregivers of Patıents with Cancer. Hemşirelikte Eğitim Ve Araştırma Dergisi, 2016;13 (3): 216-225. doi:10.5222/HEAD.2016.216.
- [Background] Yüce UÖ, Atik D, Karatepe HK, Erdoğan Z, Coşar AA. Reiki Reiki and Diabetes. Acta Med. Alanya 2017;1(2): 49-53.